CLINICAL TRIAL: NCT03057730
Title: Acellular Dermal Matrix Combined With Coronally Advanced Flap in the Treatment of Multiple Recession Defects in Thin Versus Thick Periodontal Biotype Population: A Controlled Clinical Investigation
Brief Title: A Clinical Trial Testing Root Coverage With Acellular Dermal Matrix in Thin and Thick Gingival Biotypes
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11692
Record Dates: First submitted 2017-01-18; First posted 2017-02-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Gingival Recession
Keywords: acellular dermal matrix
MeSH Terms: conditions — Gingival Recession | interventions — Alloderm

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1: Thin Biotype (Experimental): Gingival thickness < 0.8 mm
  Acellular Dermal Matrix (ADM) will be used according to manufacturer's instructions during mucogingival surgery. Subjects will be anesthetized using local anesthesia. An envelope flap design will be involved with no releasing incisions. The ADM will be placed beneath the flap. The flap will then be advanced to the level of cemento-enamel junction (CEJ). The area will be sutured.
  Mean root coverage, CPD, CAL, RH, RW, KTW, GT, and CRC will be measured and compared at 3 months, 6 months, 12 months, 24 months and 48 months post-surgery.
  Interventions: Biological: Acellular Dermal Matrix
- Group 2: Thick Biotype (Experimental): Gingival thickness ≥ 0.8 mm
  Acellular Dermal Matrix (ADM) will be used according to manufacturer's instructions during mucogingival surgery. Subjects will be anesthetized using local anesthesia. An envelope flap design will be involved with no releasing incisions. The ADM will be placed beneath the flap. The flap will then be advanced to the level of cemento-enamel junction (CEJ). The area will be sutured.
  Mean root coverage, CPD, CAL, RH, RW, KTW, GT, and CRC will be measured and compared at 3 months, 6 months, 12 months, 24 months and 48 months post-surgery.
  Interventions: Biological: Acellular Dermal Matrix

INTERVENTIONS:
Biological: Acellular Dermal Matrix — ADM is a human-derived allograft material, treated to remove all cellular components so that only the connective tissue matrix remains.
  Other Names: Alloderm®

SUMMARY:
Gingival recession is a common defect among the American population. It is also a major cause for root decay, hypersensitivity, contributes to tooth mobility and low self-esteem. Acellular dermal matrix, a human-derived grafting material has been put on the market for the treatment of gingival recession. Treating gingival recession with this material has been a validated treatment option for years.

However, treatment outcomes in two patient populations, namely those with thin biotypes and those with thick biotypes, has not been investigated. This study will observe the primary treatment outcomes in the two patient groups at 5 time points - 3 months, 6 months and 12 months post-surgery to observe short term outcomes; additional 24 months and 48 months post-surgery to observe long term outcomes.

DETAILED DESCRIPTION:
The study aim is to evaluate and compare the use of acellular dermal matrix, a material used for treating gum recession, in two study populations, namely thin or thick gingival biotype. Short term outcomes and the long term stability of ADM in recession repair between thick and thin biotypes will be evaluated.

There will be two study groups, namely thin and thick groups. The included subjects will be divided in two groups according to gingival thickness: Thin gingival biotype group (TnB): < 0.8 mm, thick gingival biotype group (TkB) ≥ 0.8 mm. Each subject will be in one of the two groups only.

Randomization will not be used to assign the subjects to the study groups, because the intervention will be the same for both groups, namely ADM applied beneath a coronally advanced flap.

The short term (3 months, 6 months post-surgery) outcomes and the longer term (12 months, 24 months and 48 months post-surgery) outcomes will further be compared within the groups and between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be current patients of Tufts University School of Dental Medicine
* Subjects with two Miller class I or class II adjacent recessions with a recession height ≥ 2 mm and < 4 mm
* Affected tooth/teeth are anterior- incisors, canines or premolars (except the mandibular central and lateral incisors)
* Healthy subjects with no contraindications to root coverage surgery
* Subjects with full-mouth plaque index<1 and gingival index<1, calculated as the average value of plaque index and gingival index

Exclusion Criteria:

* Presence of adjacent defects, whose gingival thickness values place them in a different category other than thick or thin biotype
* Areas that have previously been treated with root coverage surgeries
* Subjects with a known hypersensitivity to polysorbate 20 (contraindicated with the use of Alloderm®)
* Subject smokes more than 5 cigarettes per day
* Subjects with systemic conditions which influence wound healing
* Subjects that are pregnant or lactating
* Subjects with a condition causing immunosuppression, or currently taking immunosuppressant medications
* Teeth with severe occlusal interferences, deep cervical lesions, or large restorations whose margins impinge on the cement-enamel junction or make identification of this landmark impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change in Mean Root Coverage | Up to 48 months post surgery
  Root coverage will be measured in mm using a probe and digital caliper. Mean root coverage will be measured per patient by averaging the two study teeth. Change in mean root coverage for the primary outcome will be assessed by the difference between the baseline mean root coverage and the final mean root coverage at 48 months post surgery.

SECONDARY OUTCOMES:
Change in Clinical Probing Depth (CPD) | Up to 48 months post surgery
Change in Clinical Attachment Level (CAL) | Up to 48 months post surgery
  CAL will be measured from the base of the pocket to the cementoenamel junction (CEJ) in mm using a probe and digital caliper. Change in CAL will be assessed from baseline to 48 months post surgery.
Change in Recession Height (RH) | Up to 48 months post surgery
Change in Recession Width (RW) | Up to 48 months post surgery
Change in Keratinized Tissue Width | Up to 48 months post surgery
Change in Gingival Thickness (GT) | Up to 48 months post surgery
Complete Root Coverage (CRC) | Up to 48 months post surgery
  CRC will be assessed using descriptive statistics (# subjects with CRC out of the total sample)

CONTACTS AND LOCATIONS:
Overall Officials: Wai Cheung, DMD, MS, Principal Investigator — Tufts University School of Dental Medicine
Locations (1):
- Tufts University School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No